CLINICAL TRIAL: NCT03973476
Title: Effectiveness of Midwife Phone Support With the to Reduce the Early Abandonment of Breastfeeding
Acronym: STAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P10/53-STAM
Record Dates: First submitted 2019-04-29; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-04

CONDITIONS: Breastfeeding
Keywords: phone support; midwife; early abandonment of breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Mothers received a phone support service with their midwife during the 8 weeks after childbirth.
  Interventions: Other: Phone care support by midwife
- Control group (No Intervention): Mothers received standard postpartum care

INTERVENTIONS:
Other: Phone care support by midwife — Mothers can call the midwife's telephone every working day from 8 a.m. to 8 p.m.
  Arms: Intervention group

SUMMARY:
Objective: To evaluate the effectiveness of telephone support of the reference midwife, in relation to the abandonment of breastfeeding of primiparous mothers and to identify, both the risk factors and the protective factors for the early abandonment of breastfeeding.

Material and Method Randomized parallel controlled clinical trial.

DETAILED DESCRIPTION:
Sample: 220 primiparous mothers with access, during the 8 weeks postpartum, to a mobile phone to contact the midwife randomization of 110 mothers to the experimental group and 110 to the control group. The mothers of the experimental group will be offered the mobile phone number to contact their midwife after delivery. The mothers of the control group will receive the usual attention of the portfolio of services that includes the spontaneous visit in the center, the telephone call in the center, the home visit and the health education groups.

ELIGIBILITY:
Inclusion Criteria:

* Primiparians who carry out the follow-up of pregnancy for the midwife
* The pregnant woman is of low risk
* Possibility of the mother to make calls to the mobile phone.
* The pregnant woman wishes to participate in the study.

Exclusion Criteria

* Maternal or fetal pathology that can condition maternal breastfeeding.
* idiomatic barrier.
* Prematurity.
* Baby with weight <2,500 gr. at birth
* Home delivery during the puerperium

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who breast-feed at 3 months of intervention | 3 months
  Women who still breastfeed 3 months after the intervention with respect to the control arm

IPD SHARING:
Plan to Share IPD: No